CLINICAL TRIAL: NCT01010529
Title: Feasibility of a Trial Evaluating the Effectiveness of Occupational Therapy in Parkinson's Disease
Acronym: OTiP pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting Nuts Ohra (Other)
Responsible Party: Marten Munneke/Dr, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FNO-0804-66
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2010-10

CONDITIONS: Parkinson's Disease
Keywords: Occupational Therapy; Parkinson's Disease; Feasibility; Effectiveness; RCT; Activities of daily living; Participation; Caregiver's Burden
MeSH Terms: conditions — Parkinson Disease | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- occupational therapy (Experimental)
  Interventions: Other: occupational therapy
- No occupational therapy (No Intervention): Patients and their caregivers in the control group will have no occupational therapy intervention until their last measurement has taken place (3 months).

INTERVENTIONS:
Other: occupational therapy — Patients in the experimental group will receive 10 weeks (maximum 16 hours) occupational therapy according to a treatment protocol, which is based on the Dutch evidence based guideline for occupational therapy in Parkinson's Disease and refined for this study.
  Arms: occupational therapy

SUMMARY:
The purpose of this study is to determine the feasibility of a RCT evaluating the effectiveness of occupational therapy in Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a complex disabling condition progressively affecting activities and participation of patients. Occupational Therapy aims to optimise functional performance and engagement in meaningful roles and activities. The lack of scientific evidence for the effectiveness of Occupational Therapy (OT) in Parkinson's Disease (PD) highlights the urgent need for high quality intervention studies. The recently developed Dutch clinical practice guideline for OT in PD offers a good basis for conducting an intervention study. This proposed pilot study is an important step towards setting up a large scale RCT to evaluate the effectiveness of OT in improving daily functioning of patients with PD and reducing caregivers' burden.

ELIGIBILITY:
Inclusion criteria patients:

* idiopathic Parkinson's Disease according to UK Brain Bank Criteria
* home dwelling
* indication for occupational therapy (according to criteria in the evidence based guideline)

Inclusion criteria caregivers:

* available to provide informal support minimal two times a week to a patient who participates in the study.

Exclusion criteria patients:

* not capable of completing the self assessment forms (i.e. due to language or severe cognitive problems)
* comorbidity with symptoms that interfere with actively taking part in the intervention (e.g psychosis, severe heart condition). Or limitations in activities are dominated by the co morbid condition rather than by Parkinson's Disease.
* current participation in other allied health research (IMPACT, PARKFIT, ERGODIM)
* having received occupational therapy intervention in the last 12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Patient: Combination of AMPS-process skills and COPM-performance measure | 0 and 3 months
Caregiver: Zarit Burden Inventory (ZBI) | 0 and 3 months

SECONDARY OUTCOMES:
Patient: Assessment of Motor and Process Skills(AMPS)- motor skills | 0 and 3 months
Patient: Canadian Occupational Performance Measure (COPM)- satisfaction measure | 0 and 3 months
Patient: Impact on Participation and Autonomy (IPA) | 0 and 3 months
Patient: AMC Linear Disability Scale (ALDS) | 0 and 3 months
Patient: Parkinson's Disease Questionnaire 39 (PDQ-39) | 0 and 3 months
Patient and Caregiver: EQ-5D and VAS | 0 and 3 months
Patient and caregiver: Resource utilization | 0 and 3 months
Caregiver: Canadian Occupational Performance Measure (COPM) | 0 and 3 months
Caregiver: Questionnaire Objective Caregiving Burden | 0 and 3 months
Caregiver: SF-36 | 0 and 3 months
Patient and caregiver in intervention group: satisfaction with intervention | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Marten Munneke, Phd, Principal Investigator — UMC St Radboud
Locations (4):
- Netherlands (4):
  - Meander Medisch Centrum, locatie Elisabeth, Amersfoort
  - Gelre Ziekenhuizen, locatie Lukas, Apeldoorn
  - Alysis Zorggroep, Ziekenhuis Rijnstate, Arnhem
  - Ziekenhuis Rivierenland Tiel, Tiel